CLINICAL TRIAL: NCT05813990
Title: Reconstructive Ear Surgery in Pediatric Population. Cross Sectional Study
Brief Title: Reconstructive Ear Surgery in Pediatrics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, zeinab salah eldin mohamed, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ossiculoplasty in pediatrics
Record Dates: First submitted 2023-03-19; First posted 2023-04-14 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Ossicle Chain Disarticulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric patient with conductive hearing loss (Other): All pediatric patients aged below 18 years old will subjected to reconstructive ear surgery (ossiculoplasty)
  Interventions: Other: recostructive ear surgery

INTERVENTIONS:
Other: recostructive ear surgery — recostructive ear surgery in pediatric population
  Other Names: ossiculoplasty

SUMMARY:
The aim of the study is

1. Evaluation of preoperative degree of hearing loss in pediatric population.
2. Evaluation of types and prevalence's of ossicular disruptions due to chronic otitis media and trauma.
3. Assessment of best candidates for hearing restoration surgeries.
4. Comparing different surgical techniques for hearing restoration in various ossicular disorders .
5. Evaluation of degree of surgical restoration of the sound transmitting mechanism of the middle ear in pediatric population.

DETAILED DESCRIPTION:
Conductive hearing loss (CHL) results from impaired transmission of sound from the external auditory canal across the middle ear structures to the cochlea of the inner ear. A variety of disorders can affect the sound transmission pathway at the level of the ear canal, tympanic membrane, and ossicles prior to reaching the hearing organ.

Ossiculoplasty is the surgical restoration of the sound transmitting mechanism of the middle ear. Ossiculoplasty has been performed as early as the 1950s.A myriad of prosthetics and surgical techniques have been described over the last half-century, with no overall consensus on the ideal method of treatment.

Pediatric population are commonly known to develop conductive hearing loss secondary to various conditions such as chronic otitis media, otitis media with effusion, atelectatic otitis media and head trauma. Various methods have been fashioned to restore hearing in such patients however no consensus to the most optimum method for hearing restoration has been well established

ELIGIBILITY:
Inclusion Criteria:

1. patients aged ≤ 18years with CHL.
2. patients who are candidate for ossiculoplasty as surgical treatment for them.

Exclusion Criteria:

1. Patients with preoperative sensory neural hearing loss (SNHL).
2. Patient with intra operative complications.
3. Patients with intracranial and intratemporal complications.
4. Patients with stapes foot plate fixation, broken graft and missed patients.
5. Patients >18years.
6. Patients who unfit for surgery.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
reconstuctive ear surgery in pediartic population | 2m,6m and 1year
  Evaluation of degree of surgical restoration of the sound transmitting mechanism of the middle ear in pediatric population using audiometry 2 months, 6month and 1 year after surgery to assess hearing results and prosthesis stability.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

REFERENCES:
- [Background] Kamrava B, Roehm PC. Systematic Review of Ossicular Chain Anatomy: Strategic Planning for Development of Novel Middle Ear Prostheses. Otolaryngol Head Neck Surg. 2017 Aug;157(2):190-200. doi: 10.1177/0194599817701717. Epub 2017 May 2. PMID 28463590